CLINICAL TRIAL: NCT02271373
Title: Development and Application of Appropriate Technology for Myopia Prevention and Control
Brief Title: Effect of Increasing Time Spent Outdoors on Myopia Prevention in School-Aged Children in Northeast China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Fangbiao Tao, Dean of School of Public Health, Anhui Medical University, Anhui Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013001
Record Dates: First submitted 2014-10-19; First posted 2014-10-22 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Myopia
Keywords: Vision, Ocular; Physical activity; Schoolchildren; Intervention Studies
MeSH Terms: conditions — Myopia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): The intervention group undertook interventions by increasing time spent outdoors. The interventions composed of performing two additional recess program lasting 30 minutes outside the classroom that encouraged children to go outside for outdoor activities during recess in both the morning and afternoon during school days within a intervention period of 1 school year.
  Interventions: Behavioral: increasing time spent outdoors
- control group (No Intervention): The control school did not have any interventions.

INTERVENTIONS:
Behavioral: increasing time spent outdoors — The intervention group undertook interventions by increasing time spent outdoors. The interventions composed of performing two additional recess program lasting 30 minutes outside the classroom that encouraged children to go outside for outdoor activities during recess in both the morning and afternoon during school days within a intervention period of 1 school year.
  Arms: intervention group

SUMMARY:
The purpose of this study is to develop a school-based intervention aimed at prevent the onset and development of myopia among school aged children by increasing time spent outdoors in northeast China.

DETAILED DESCRIPTION:
The purpose of this study is to develop a school-based intervention aimed at prevent the onset and development of myopia among school aged children by increasing time spent outdoors among elementary and secondary school students in northeast China. It is expected that the results will provide evidences for policy-makers and school healthcare providers for their school children myopia prevention.

ELIGIBILITY:
Inclusion Criteria:

* Grade of 1 to 5 in elementary schools and grade of 7 to 8 in secondary schools.

Exclusion Criteria:

* Visual defect or other eye diseases; wearing orthokeratology; refractive surgery history.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3521 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes in uncorrected visual acuity | Baseline, Month 6, Month 12
  Uncorrected visual acuity (UCVA) was measured for the right eye, then the left eye, with a E Standard Logarithm Vision Acuity Chart (GB11533-2011) in 5-grade notation (5- LogMAR), with illumination of the chart around 500lx. If one of the eyes UCVA was less than 5.0, then tests with combined lenses were conducted among the poor eye-sighted for confirming the types of ametropia (normal, myopia, hyperopia or other eye diseases)．All the measurements were recorded.

SECONDARY OUTCOMES:
Questionnaire survey | Baseline
  The parents and children underwent an interview together. The questionnaire included questions on children's gender, ethnicity, region of habitation; questions on parental education level, the monthly family income and whether the parents were myopic or not;. The interview also included questions on the amount of time spent for learning (reading or writing), screen time (television, computer, etc) and time spent outdoors after school in recent 7 days.
Changes in ocular biometric parameters | Baseline, Month 12
  A random subsample (12.8%) underwent cycloplegia. After ensuring that there was no risk for a medical mydriasis, cycloplegia was performed at baseline and intervention after 1 year in the Shenyang Aier Ophthalmology Hospital, respectively. Ocular biometric parameters (axial length, corneal curvature, anterior chamber depth and IOP) were measured in both eyes of all participants. Axial length, corneal curvature and anterior chamber depth were measured with IOL Master (intraoeular len master, IOL. Master) (Carl Zeiss Meditex, Jena, Germany); Intraocular pressure (IOP) measurement was obtained using a non-contact tonometry (NT-510, NIDEK, Gamagori, Japan). Cycloplegia was achieved by 0.5% tropicamide eye drops. Six drops of tropicamide 0.5% were administered at 5-minute intervals for both eyes. Refractometry was performed 20 minutes after the last cycle of cycloplegic eye drops by retinoscopy (YZ-24, Suzhou, China).

CONTACTS AND LOCATIONS:
Overall Officials: Fangbiao Tao, PhD, Study Director — Department of Maternal, Child and Maternal Health, School of Public Health, Anhui Medical University

REFERENCES:
- [Derived] Jin JX, Hua WJ, Jiang X, Wu XY, Yang JW, Gao GP, Fang Y, Pei CL, Wang S, Zhang JZ, Tao LM, Tao FB. Effect of outdoor activity on myopia onset and progression in school-aged children in northeast China: the Sujiatun Eye Care Study. BMC Ophthalmol. 2015 Jul 9;15:73. doi: 10.1186/s12886-015-0052-9. PMID 26152123